CLINICAL TRIAL: NCT00933933
Title: Evaluation of ARCHITECT HIV Ag/Ab Combo Assay
Brief Title: Evaluation of Diagnostic HIV Ag/Ab Combo Assay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Barbara Kaesdorf, Clinical Project Manager, Abbott Diagnostics Division
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7B5-02-06R01
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2010-08-19 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Human Immunodeficiency Viruses
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARCHITECT HIV Ag/Ab Combo Specificity (Experimental): Specimens collected from normal apparently healthy individuals at low risk for HIV infection will be tested by the investigational HIV test and FDA-licensed HIV test.
  Interventions: Device: ARCHITECT HIV Ag/Ab Combo
- ARCHITECT HIV Ag/Ab Combo Sensitivity (No Intervention): Specimen with confirmed positive HIV Antigen, HIV-1 antibody, or HIV-2 antibody will be tested by the investigational HIV test.
- ARCHITECT HIV Ag/Ab Combo Reactivity (Experimental): Specimen collected from individuals at risk for HIV infection will be tested by the investigational HIV test.
  Interventions: Device: ARCHITECT HIV Ag/Ab Combo

INTERVENTIONS:
Device: ARCHITECT HIV Ag/Ab Combo — Test blood samples with investigational HIV assay. If results for specimens from the normal healthy population or pregnant female population at risk for HIV infection are reactive, samples will be tested with supplemental HIV assays. If all supplemental HIV assays are negative, subject will be asked to return for a follow-up blood draw.
  Arms: ARCHITECT HIV Ag/Ab Combo Specificity
Device: ARCHITECT HIV Ag/Ab Combo — Test blood samples with investigational HIV assay. If results for specimens from the at risk population are reactive, samples will be tested with supplemental HIV assays. If all supplemental HIV assays are negative, subject will be asked to return for a follow-up blood draw when possible.
  Arms: ARCHITECT HIV Ag/Ab Combo Reactivity

SUMMARY:
To test blood specimens using a new investigational test that detects antigen and antibody to human immunodeficiency virus (HIV). Results will be compared to an approved HIV antibody test and supplemental testing performed to determine HIV status.

DETAILED DESCRIPTION:
All specimens collected under separate specimen collection protocols or obtained from specimen suppliers will be provided to the clinical sites performing the investigational HIV test.

This includes 6252 specimens collected from normal healthy individuals (7B5-02-05Z01-01: Collection of Specimens Used in Abbott Laboratories In Vitro Diagnostic HIV and Hepatitis Assays Clinical Studies)and from specimen suppliers. 588 specimens from HIV-infected pediatric subjects and 448 pregnant females at risk for HIV infection collected under protocol (7B5-02-05Z01-02: Collection of Pediatric and Pregnant Female Specimens Used in the Abbott Laboratories In Vitro Diagnostic HIV Assay)and from specimen suppliers. All specimens were previously collected and frozen, except for a subset of 586 specimens from normal healthy population and 55 specimen from pregnant females at risk for HIV infection which were collected under separate specimen collection protocols and tested as fresh specimens during the study.

In addition, 83 specimens that were HIV antigen positive, 1121 specimens that were HIV-1 antibody positive, 201 specimens that were HIV-2 antibody positive, and 1409 specimens from US at risk for HIV infection or from HIV-2 endemic area were all obtained from specimen suppliers, except for 11 pediatric specimens collected under a separate protocol (7B5-02-05Z01-02: Collection of Pediatric and Pregnant Female Specimens Used in the Abbott Laboratories In Vitro Diagnostic HIV Assay).

ELIGIBILITY:
Normal Healthy Population:

Inclusion Criteria:

* Apparently healthy individual at the time of enrollment as affirmed by the subject

Exclusion Criteria:

* HIV infection as affirmed by the subject

Pregnant Female Population at Risk for HIV Infection:

Inclusion Criteria:

* Subject is a pregnant female
* Subject has risk factor for HIV infection

Exclusion Criteria:

* HIV infection as affirmed by the subject

HIV-1 Positive Pregnant Female Subjects

Inclusion Criteria:

* Subject is a pregnant female in first, second, or third trimester
* Subject must have documented HIV infection

Exclusion Criteria:

* None

HIV-1 Positive Pediatric Subjects

Inclusion Criteria:

* Subject must be 2 years to 16 years of age
* Subject must have documented HIV infection (e.g., Western blot positive or HIV RNA positive/detectable)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Roberts, MD, Principal Investigator — ARUP Laboratories; Laurence Demers, PhD, Principal Investigator — M.S. Hershey Medical Center; Fred Apple, PhD, Principal Investigator — Hennepin Healthcare Research Institute; Michael Loeffelholz, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston; John Heffner, Principal Investigator — Clement J. Zablocki VA Medical Center
Locations (13):
- United States (13):
  - Radiant Research, Phoenix, Arizona
  - Pinellas County Health Dept, Florida Department of Health, St. Petersburg, Florida
  - Springfield Clinic, LLP, Springfield, Illinois
  - Minneapolis Medical Research Foundation, Minneapolis, Minnesota
  - John T. Mather Memorial Hospital, Port Jefferson, New York
  - Jacobi Medical Center, The Bronx, New York
  - M.S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Planned Parenthood of Houston and Southeast Texas, Inc., Houston, Texas
  - ARUP Laboratories, Salt Lake City, Utah
  - Midwest Research Specialists, LLC, Milwaukee, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All specimens collected under separate collection protocols or obtained from specimen suppliers: human immunodeficiency virus (HIV) antigen positive samples, HIV-1 antibody positive, specimens collected from individuals at risk for HIV infection in the United States (US), HIV-2 antibody positive and specimens collected from HIV-2 endemic area.
Pre-assignment Details: All subjects were assigned to one group. There was no pre-screening criteria for this study.
Groups:
- Architect HIV Ag/Ab Combo Specificity: Specificity populations included:
  6164 specimens collected from apparently healthy individuals at low risk for HIV infection (16-89 years of age) which includes 250 specimens from pregnant females in first trimester of pregnancy.
  448 specimen from presumed HIV negative pregnant females from 16 to 44 years of age.
  588 specimen from pediatric presumed negative for HIV from 2 to 21 years of age.
  Specimens were collected under separate collection protocols or by specimens vendors and tested with investigation HIV test.
- Architect HIV Ag/Ab Combo Sensitivity: Sensitivity populations included:
  1287 specimens or commercial panel members HIV-1 p24 Antigen positive, specimens confirmed HIV-1 antibody positive and specimens confirmed HIV-2 antibody positive.
  67 specimens from pregnant females from all three trimesters confirmed HIV posiitve by supplemental testing.
  64 specimens from pediatric subjects confirmed HIV positive by supplemental testing (2 to 21 years of age).
  Specimens were collected under separate collection protocols or by specimens vendors and tested with investigational HIV test.
- Architect HIV Ag/Ab Combo Reactivity: Reactivty populations included:
  1206 specimens collected from individuals at increased risk for HIV infection (16-89 years of age) from US and Cote D'Ivoire.
  203 specimen from pregnant females at risk for HIV infection.
  Of these 1409 specimens, 61 were collected from individual that were from 16 up to 21 years of age.
  Specimens were collected under separate collection protocols or by specimens vendors and tested with investigation HIV test.
Period: General Population From 16 to 89 Years
Arm/Group | Architect HIV Ag/Ab Combo Specificity | Architect HIV Ag/Ab Combo Sensitivity | Architect HIV Ag/Ab Combo Reactivity
Started | 6164 | 1287 | 1206
Completed | 6164 | 1267 | 1206
Not Completed | 0 | 20 | 0
Not completed — Did not meet criteria for analysis | 0 | 20 | 0
Period: Pregnant Females Between 16-44 Years
Arm/Group | Architect HIV Ag/Ab Combo Specificity | Architect HIV Ag/Ab Combo Sensitivity | Architect HIV Ag/Ab Combo Reactivity
Started | 448 | 67 | 203
Completed | 448 | 65 | 203
Not Completed | 0 | 2 | 0
Not completed — Specimens classified incorrectly | 0 | 2 | 0
Period: Pediatric From 2 to 21 Years
Arm/Group | Architect HIV Ag/Ab Combo Specificity | Architect HIV Ag/Ab Combo Sensitivity | Architect HIV Ag/Ab Combo Reactivity
Started | 588 | 64 | 0 (Specimens from individuals 16-21 years included reactivity for general population or pregnant women.)
Completed | 588 | 64 | 0 (Specimens from individuals 16-21 years included reactivity for general population or pregnant women)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Architect HIV Ag/Ab Combo Specificity: Specimens collected from apparently healthy individuals under a separate specimen collection protocol (7B5-02-05Z01-01) or obtained from specimen vendors and were tested with investigational HIV test.
- Architect HIV Ag/Ab Combo HIV-1 Antigen Sensitivity; Architect HIV Ag/Ab Combo HIV-2 Antibody Sensitivity: Specimens obtained from specimen vendors were tested with investigational HIV test.
- Architect Ag/Ab Combo HIV-1 Antibody Sensitivity: Specimens collected from HIV-1 infected individuals under a separate specimen collection protocol (pediatric subjects 7B5-02-05Z01-02) or obtained from specimen vendors and were tested with investigational HIV test.
- Architect HIV Ag/Ab Combo Reactivity: Specimens collected from individuals at increased risk for HIV infection under a separate specimen collection protocol (pregant females 7B5-02-05Z01-02) or obtained from specimen vendors and were tested with investigational HIV test.
- Total: Total of all reporting groups
Arm/Group | Architect HIV Ag/Ab Combo Specificity | Architect HIV Ag/Ab Combo HIV-1 Antigen Sensitivity | Architect Ag/Ab Combo HIV-1 Antibody Sensitivity | Architect HIV Ag/Ab Combo HIV-2 Antibody Sensitivity | Architect HIV Ag/Ab Combo Reactivity | Total
Number analyzed (Participants) | 6252 | 83 | 1121 | 201 | 1409 | 9066
Age, Customized [Number; unit: participants]
  between 2 and 21 years | 588 | 0 | 64 | 0 | 61 | 713
  >= 21 years | 5663 | 0 | 1057 | 0 | 1304 | 8024
  Not collected | 1 | 83 | 0 | 201 | 44 | 329
Sex/Gender, Customized [Number; unit: participants]
  Female | 4165 | 0 | 231 | 0 | 530 | 4926
  Male | 2087 | 0 | 890 | 0 | 879 | 3856
  Not collected | 0 | 83 | 0 | 201 | 0 | 284
Region of Enrollment [Number; unit: Participants]
  United States | 6252 | 78 | 1121 | 0 | 896 | 8347
  Côte D'Ivoire | 0 | 0 | 0 | 201 | 513 | 714
  South Africa | 0 | 4 | 0 | 0 | 0 | 4
  Cameroon | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Architect HIV Combo Test Data for Clinical Specificity in Population at Low Risk for HIV Infection
Description: HIV status was determined by the results of the HIV comparator assay, HIV-1 Western blot, HIV-2 Western blot, and HIV-1 ribonucleic acid (RNA) test.
Time Frame: 3 months
Population: Specificity determined from 6,164 specimens from apparently healthy individuals (low risk): includes 250 specimens from pregnant females in first trimester and 580 specimens from low risk population prospectively collected and tested fresh during study. Total of 37 confirmed HIV positives by supplemental testing were excluded from analysis.
Measure: Number; unit: Blood Specimens
Groups:
- Architect HIV Ag/Ab Specificity - Low Risk for HIV Infection: Specimens collected from a population of apparently healthy individuals at low risk for HIV infection.
Arm/Group | Architect HIV Ag/Ab Specificity - Low Risk for HIV Infection
Number analyzed (Participants) | 6164
Blood Specimens
  HIV Ag/Ab Combo Reactive, HIV status Positive | 37 [99.62 to 99.88]
  HIV Ag/Ab Combo Reactive, HIV status Negative | 14
  HIV Ag/Ab Combo Nonreactive HIV status Positive | 0
  HIV Ag/Ab Combo Nonreactive HIV status Negative | 6113
Statistical Analysis 1: Comparison: Architect HIV Ag/Ab Specificity - Low Risk for HIV Infection; Test type: Superiority or Other; Exact binomial; Clinical Specificity = 99.77, 95% CI 2-sided [99.62 to 99.88]

2. Primary Outcome: Architect HIV Combo Test Data for Clinical Sensitivity in HIV Positive Specimens
Description: Positive HIV status was determined by the results of the HIV-1 Western blot, HIV-2 Western blot, and/or HIV-1 ribonucleic acid (RNA) test.
Time Frame: 3 months
Population: Sensitivity was determine using confirmed positive specimens/panels for HIV-1 Antigen (63 samples/panels/viral isolates), HIV-1 antibody (1003 US population) and HIV-2 antibody (201 endemic area of Ivory Coast) based on supplemental testing.
Measure: Number; unit: Blood specimens
Groups:
- HIV p24 Antgen Sensitivity: HIV-1 Antigen positive specimens/commercial panel members (HIV Westerm blot negative and confirmed positive by HIV-1 p24 Antigen and/or HIV RNA) and HIV-1 viral isolates.
- HIV-1 Antibody Sensitivity: Specimens collected from HIV infected individuals in US population confirmed by HIV-1 Western blot.
- HIV-2 Antibody Sensitivity: Specimens collected from HIV infected individuals in Ivory Coast confirmed by HIV-2 Western blot.
Arm/Group | HIV p24 Antgen Sensitivity | HIV-1 Antibody Sensitivity | HIV-2 Antibody Sensitivity
Number analyzed (Participants) | 63 | 1003 | 201
Blood specimens
  ARCHITECT HIV Ag/Ab Reactive | 63 | 1003 | 201
  ARCHITECT HIV Ag/Ab Nonreactive | 0 | 0 | 0
Statistical Analysis 1: Comparison: HIV p24 Antgen Sensitivity; Test type: Superiority or Other; Exact binomial; Clinical Sensitivity = 100.00, 95% CI 2-sided [94.31 to 100.00]
Statistical Analysis 2: Comparison: HIV-1 Antibody Sensitivity; Test type: Superiority or Other; Exact binomial; Clinical Sensitivity = 100.00, 95% CI 2-sided [99.63 to 100.00]
Statistical Analysis 3: Comparison: HIV-2 Antibody Sensitivity; Test type: Superiority or Other; Exact binomial; Clinical Sensitivity = 100.00, 95% CI 2-sided [98.18 to 100.00]

3. Primary Outcome: Architect HIV Combo Test Data for Specificity and Sensitivity in Pregnant Female Population
Description: as for outcome 1
Time Frame: 3 months
Population: HIV negative status determined for specimens reactive by investigational assay and/or comparator by supplemental testing algorithm including HIV-1 Western blot, HIV-2 enzyme immunoassay (EIA), HIV-2 Western blot, HIV-1 p24 Antigen assay and HIV-1 RNA. HIV positive status determined by HIV-1 Western blot. Specimens from pregnant females.
Measure: Number; unit: Blood specimens
Groups:
- Architect HIV Ag/Ab Combo Specificity in Pregnant Females: HIV presumed negative specimens from pregnant females tested with investigation HIV test, comparator assay and supplemental tests.
- Architect HIV Ag/Ab Combo Sensitivity in Pregnant Females: HIV confirmed positive specimens from pregnant females tested with investigation HIV test, comparator assay and supplement tests.
Arm/Group | Architect HIV Ag/Ab Combo Specificity in Pregnant Females | Architect HIV Ag/Ab Combo Sensitivity in Pregnant Females
Number analyzed (Participants) | 448 | 65
Blood specimens
  Architect HIV Ag/Ab Reactive | 0 | 65
  Architect HIV Ag/Ab Nonreactive | 448 | 0
Statistical Analysis 1: Comparison: Architect HIV Ag/Ab Combo Specificity in Pregnant Females; Test type: Superiority or Other; Exact binomial; Clinical Specificity = 100.00, 95% CI 2-sided [99.18 to 100.00]
Statistical Analysis 2: Comparison: Architect HIV Ag/Ab Combo Sensitivity in Pregnant Females; Test type: Superiority or Other; Exact binomial; Clinical Sensitivity = 100.00, 95% CI 2-sided [94.48 to 100.00]

4. Primary Outcome: Architect HIV Combo Test Data for Specificity and Sensitivity in Pediatric Population (From 2 up to 21 Years of Age)
Description: as for outcome 1
Time Frame: 3 months
Population: Specificity determine from 588 specimens: 364 low risk, 95 increased risk, 47 increased risk (HIV-2 endemic area), 44 pregnant females low risk and 38 pregnant females increased risk with HIV negative status. Sensitivity determined from 65 specimens: 60 HIV-1 infected, 2 HIV-1 infected pregnant females, 2 HIV infected from HIV-2 endemic area.
Measure: Number; unit: Blood specimens
Groups:
- Architect HIV Ag/Ab Combo Specificity in Pediatric Population: Specimens presumed HIV negative tested with investigational HIV test, FDA-licensed comparator assay and supplemental tests. Specimens from individuals between 2 and 21 years of age.
- Architect HIV Ag/Ab Combo Sensitivity in Pediatric Population: Specimens confirmed HIV positive by HIV-1 Western blot were tested with investigational HIV test. Specimens from individuals between 2 and 21 years of age.
Arm/Group | Architect HIV Ag/Ab Combo Specificity in Pediatric Population | Architect HIV Ag/Ab Combo Sensitivity in Pediatric Population
Number analyzed (Participants) | 588 | 64
Blood specimens
  HIV Ag/Ab Combo Reactive HIV Status Positive | 0 | 64
  HIV Ag/Ab Combo Reactive HIV Status Negative | 1 | 0
  HIV Ag/Ab Combo Nonreactive HIV Status Positive | 0 | 0
  HIV Ag/Ab Combo Nonreactive HIV Status Negative | 587 | 0
Statistical Analysis 1: Comparison: Architect HIV Ag/Ab Combo Specificity in Pediatric Population; Test type: Superiority or Other; Exact binomial; Clinical Specificity = 99.83, 95% CI 2-sided [99.06 to 100.00]
Statistical Analysis 2: Comparison: Architect HIV Ag/Ab Combo Sensitivity in Pediatric Population; Test type: Superiority or Other; Exact binomial; Clinical Sensitivity = 100.00, 95% CI 2-sided [94.40 to 100.00]

5. Secondary Outcome: Architect HIV Combo Test Data for Reactivity of Architect HIV Combo in Increased HIV Risk Populations
Description: Reactivity was determined by the results of the Architect HIV Ag/Ab Combo assay and supplemental testing by HIV-1 Western blot, HIV-2 Western blot, and HIV-1 ribonucleic acid (RNA) test.
Time Frame: 3 months
Population: Final HIV status determined for specimens reactive by investigational assay and/or comparator by supplement testing algorithm. Supplemental testing involved HIV-1 Western blot, HIV-2 EIA, HIV-2 Western blot, HIV-1 p24 Antigen assay and HIV-1 RNA. HIV positive status determined by HIV-1 Western blot.
Measure: Number; unit: Blood specimens
Groups:
- Increased Risk for HIV in US Population: Specimens collected from 693 individuals in the US population documented as having one or more of the following risk factors: users of injecting drugs, unprotected sex with someone who is infected with HIV, diagnosed or treated for a sexually transmitted disease (STD), hepatitis or tuberculosis, multiple sex partners, men who have sex with men, men who have sex with men and are users of injecting drugs, unprotected sex with someone who has been diagnosed or treated for an STD, risk factor not identified but requested an HIV test. Specimens obtained from specimen vendors and were tested with investigational HIV test.
- Increased Risk for HIV From HIV-2 Endemic Area: Specimens from 513 individuals documented as being at risk for acquiring HIV that reside in an HIV-2 endemic area (Cote De'Ivoire) having one or more of the following risk factors: unprotected sex with someone who is infected with HIV, multiple sex partners, men who have sex with men, users of injecting drugs. Specimens were obtained from specimen vendors and tested with investigational HIV test.
- Reactivity in Pregnant Female Population: Specimens collected from 203 pregnant females: 153 specimens collected from pregnant females with documented risk factors for HIV and 50 were surplus serum specimens collected pregnant females from a health clinic offering HIV testing. Spcimens from 55 of the pregnant females with risk for HIV infection were collected under a specimen collection protocol and tested with the investigational and FDA-licensed comparator assay during the study. The remaining specimens were obtained from specimen vendors and tested with the investigational HIV test.
Arm/Group | Increased Risk for HIV in US Population | Increased Risk for HIV From HIV-2 Endemic Area | Reactivity in Pregnant Female Population
Number analyzed (Participants) | 693 | 513 | 203
Blood specimens
  HIV Ag/Ab Combo Reactive HIV Status Positive | 65 | 83 | 5
  HIV Ag/Ab Combo Reactive HIV Status Negative | 6 | 6 | 0
  HIV Ag/Ab Combo Nonreactive - HIV Status Positive | 0 | 0 | 0
  HIV Ag/Ab Combo Nonreactive HIV Status Negative | 622 | 424 | 198

ADVERSE EVENTS:
Time Frame: Device adverse events were collected during the approximate 3 months of testing with Architect HIV Combo assay.
Description: Adverse event reporting for follow-up collection (3) and subject's with specimens collected/tested during study (635)were under separate specimens collection protocol. Not applicable for specimens collected and banked or obtained from specimen venders and provided to testing site by Abbott.
Groups:
- Architect HIV Ag/Ab Combo Specificity; Architect HIV Ag/Ab Combo Sensitivity; Architect HIV Ag/Ab Combo Reactivity: Specimens collected from specimen vendors or from specimen collection studies were tested with investigation HIV test.
Arm/Group | Architect HIV Ag/Ab Combo Specificity | Architect HIV Ag/Ab Combo Sensitivity | Architect HIV Ag/Ab Combo Reactivity
Serious Adverse Events (participants affected / at risk) | 0/586 | 0/0 | 0/55
Other Adverse Events (participants affected / at risk) | 0/586 | 0/0 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) must provide copy of any proposed publication/presentation at least 30 days prior to submission for sponsor review/approval. PI must incorporate changes as the sponosr requires in order to protect the sponsor's proprietary rights and interests. Sponsor may require the PI to include acknowledgement of sponosr's role in the study. PI may be requested to delay publication/presentation an extra 60 days to enable sponor to secure patent or other proprietary protection.